CLINICAL TRIAL: NCT05275114
Title: Improvement Effect of Transcranial Direct Current Stimulation (tDCS) Applied During Exercise Training in Stroke Patients With Upper Limb and Hand Motor Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yun-Hee Kim (Other)
Collaborators: Cybermedic Co., Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, Yun-Hee Kim, Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-06-176
Record Dates: First submitted 2022-03-01; First posted 2022-03-11 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand Tasks + M1(1mA) & aIPS(1mA) tDCS (Experimental): 20 minutes of Hand Taks + applying 30 minutes of M1(1mA) & aIPS(1mA) tDCS and fNIRS
  Interventions: Device: tDCS stimulation with hand task
- Hand Tasks + Sham tDCS (Active Comparator): 20 minutes of Hand Tasks + 30 minutes of sham tDCS and fNIRS
  Interventions: Device: sham tDCS stimulation with hand task

INTERVENTIONS:
Device: tDCS stimulation with hand task — 30 minutes of intervention including tDCS stimulation with hand task and fNIRS measurements for 10 days in 4 weeks
  Arms: Hand Tasks + M1(1mA) & aIPS(1mA) tDCS
Device: sham tDCS stimulation with hand task — 30 minutes of intervention including sham tDCS stimulation with hand task and fNIRS measurements for 10 days in 4 weeks
  Arms: Hand Tasks + Sham tDCS

SUMMARY:
The purpose of this study was to improve the effect of Transcranial Direct Current Stimulation (tDCS) applied during exercise training in stroke patients with upper limb and hand motor function.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 to 80 years
* Less than 58 FMA Upper scores
* Patients whose lesions do not include stimulation regions
* Patients with stroke with more than 3 months of onset

Exclusion Criteria:

* Difficult to communicate due to severe language impairment.
* Accompanied by an existing serious neurogenic disease
* Existing significant psychiatric disorders such as major schizophrenia, bipolar disorder
* If there are difficulties in conducting the research
* Any patients who are judged by the investigator to be difficult to participate in this study
* Patients with contraindicated MRI scans

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Assessment | Session 0 (initial visit);; Session 10 (at approximatel 4 weeks)
  The score is a stroke-specific, performance-based impairment index. The degree of impairment of upper and lower limbs is measured.

SECONDARY OUTCOMES:
Change in 9-hole pegboard test | Baseline(initial visit); Session 10 (at approximatel 4 weeks)
  The test is a standardized, quantitative assessment used to measure finger dexterity of a patient.
Change in Grip & Tip pinch strength | Baseline(initial visit); Session 10 (at approximatel 4 weeks)
  The test is to measure the maximum isometric strength of hand, forearm, and finger muscles.
Change in Sequential finger tapping reaction time and accruacy | Baseline(initial visit); Session 10 (at approximatel 4 weeks)
  Response time and accuracy are measured during finger tapping task.
Change in Jebsen-Taylor hand function test | Baseline(initial visit); Session 10 (at approximatel 4 weeks)
  This test is a standardized and objective measure of fine and gross motor hand function using simulated activities of daily living (ADL).
Change in Box and Block test | Baseline(initial visit); Session 10 (at approximatel 4 weeks)
  The test is used to measure the gross manual dexterity of a patient, or of a person using an upper limb prosthetic device.
Changes in motor evoked potential | [Time Frame: session 0 (initial visit); session 10 (at approximately 4 weeks)]
  Resting motor threshold (rMT) and amplitude of motor evoked potential in first dorsal interosseous muscle are measured. These outcomes are measured by transcranial magnetic stimulation over the motor hotspot. The rMT is defined as the minimum stimulus intensity that produced a minimal motor evoked response at rest. The amplitude means peak to peak of the muscle response.
Changes in Brain activation of resting-state functional MRI | [Time Frame: session 0 (initial visit); session 10 (at approximately 4 weeks)]
  Measure of Neuroplasticity

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lee SH, Lee G, Kim J, Phillips V Z, Kim H, Kim E, Lee SH, Jeong HC, Paik SH, Kim YH, Kim BM. Resting-state hemodynamic changes and effects on upper limb function after multi-channel transcranial direct current stimulation to the ipsilesional primary motor cortex and anterior intraparietal sulcus in stroke patients: an fNIRS pilot study. J Neuroeng Rehabil. 2025 Apr 16;22(1):83. doi: 10.1186/s12984-025-01618-8. PMID 40241110